CLINICAL TRIAL: NCT03056755
Title: BYLieve: A Phase II, Multicenter, Open-label, Three-cohort, Non- Comparative Study to Assess the Efficacy and Safety of Alpelisib Plus Fulvestrant or Letrozole in Patients With PIK3CA Mutant, Hormone Receptor (HR) Positive, HER2-negative Advanced Breast Cancer (aBC), Who Have Progressed on or After Prior Treatments
Brief Title: Study Assessing the Efficacy and Safety of Alpelisib Plus Fulvestrant or Letrozole, Based on Prior Endocrine Therapy, in Patients With PIK3CA Mutant, HR+, HER2- Advanced Breast Cancer Who Have Progressed on or After Prior Treatments
Acronym: BYLieve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X2402; 2023-509167-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: advanced breast cancer; PIK3CA; CDK 4/6 inhibitor; fulvestrant; letrozole; HR+; HER2-negative; post menopausal; pre-menopausal; aromatase inhibitor; endocrine treatment; AI; ET
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib; Fulvestrant; Letrozole; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Pre-treated with CDK 4/6i + AI (Experimental): Participants who received any Cyclin-Dependent Kinases 4 and 6 inhibitor (CDK 4/6i) plus aromatase inhibitor (AI) as immediate prior treatment will receive alpelisib + fulvestrant
  Interventions: Drug: Alpelisib; Drug: Fulvestrant; Drug: Goserelin; Drug: Leuprolide
- Cohort B: Pre-treated with CDK 4/6i + fulvestrant (Experimental): Patients who received any CDK 4/6i plus fulvestrant as immediate prior treatment will receive alpelisib + letrozole
  Interventions: Drug: Alpelisib; Drug: Letrozole; Drug: Goserelin; Drug: Leuprolide
- Cohort C: Pre-treated with systemic chemotherapy or ET (Experimental): Participants who received systemic chemotherapy or endocrine therapy (ET) (as monotherapy or in combination with targeted treatment except CDK 4/6i + AI) as immediate prior treatment will receive alpelisib + fulvestrant.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant; Drug: Goserelin; Drug: Leuprolide

INTERVENTIONS:
Drug: Alpelisib — 300 mg of alpelisib film-coated tablets administered orally once daily
  Other Names: BYL719
Drug: Fulvestrant — 500 mg of fulvestrant via intramuscular injection administered on Days 1, 15 on Cycle 1 and Day 1 at each cycle thereafter. Cycle=28 days
  Arms: Cohort A: Pre-treated with CDK 4/6i + AI; Cohort C: Pre-treated with systemic chemotherapy or ET
Drug: Letrozole — 2.5 mg of letrozole film-coated tablets administered orally once daily
  Arms: Cohort B: Pre-treated with CDK 4/6i + fulvestrant
Drug: Goserelin — 3.6 mg of goserelin via injectable subcutaneous implant administered every 28 days. Only for men in Cohort B and premenopausal women.
Drug: Leuprolide — 7.5 mg of leuprolide via injectable intramuscular depot administered every 28 days. Only for men in cohort B and premenopausal women.

SUMMARY:
This was a Phase II, multicenter, open-label, three-cohort, non-comparative study of alpelisib plus endocrine therapy (either fulvestrant or letrozole) in subjects (pre- and post-menopausal women and men) with HR-positive, HER2-negative aBC harboring PIK3CA mutation(s) in the tumor, whose disease had progressed on or after prior treatments.

DETAILED DESCRIPTION:
The study comprised two phases:

1. Core Phase: included a treatment phase for all subjects from first subject first treatment (FSFT) until disease progression, unacceptable toxicity, or death until 18 months post last subject first treatment (LSFT) + 1 month safety follow-up (total 19 months post LSFT), discontinuation from the study treatment for any other reason, or sponsor terminates the study. At the start of the Core Phase, subjects were assigned to Cohort A, Cohort B, or Cohort C based on previous therapy as follows:

   * Cohort A: alpelisib (300 mg oral QD) + fulvestrant (500 mg intramuscular (IM)) to subjects whose last prior treatment was a CDK4/6i plus any AI;
   * Cohort B: alpelisib (300 mg oral QD) + letrozole (2.5 mg oral QD) to subjects whose last prior treatment was a CDK4/6i plus fulvestrant;
   * Cohort C: alpelisib (300 mg oral QD)+ fulvestrant (500 mg IM) to subjects who failed prior AI based therapy and whose last prior treatment was systemic chemotherapy or endocrine therapy (as monotherapy or in combination with targeted treatment except CDK 4/6i + AI). Endocrine therapy included letrozole, fulvestrant and CDK 4/6 inhibitor plus fulvestrant.
2. Extension Phase: included a treatment phase starting at the end of the treatment Core Phase until last subject last visit(LSLV) (up to 36 months). Following the end of the Core Phase, subjects continuing to derive benefit from study treatment who were not eligible for Post-Study Drug Supply (PSDS) in their country based on local regulations were re-consented and transitioned to the Extension Phase. Subjects continued on their existing study treatment assigned in the Core Phase until disease progression/lack of clinical benefit or any other reason for which the subject may have been discontinued from study treatment. If PSDS became available for a subject, the subject was to be discontinued from the study and to access treatment via PSDS. When subjects discontinued treatment for any reason, the end of treatment visit was performed after discontinuation of the medication , followed by safety follow-up 30 days after last dose.

A total of 340 subjects were planned to be enrolled, with approximately 112 subjects in each cohort. In the Core Phase, 379 subjects were analyzed, with 127 subjects in Cohort A, 126 subjects in Cohort B, and 126 subjects in Cohort C. In the Extension Phase, 11 subjects were analyzed, with 1 subject in Cohort A and 10 subjects in Cohort C.

ELIGIBILITY:
Key Inclusion Criteria: Subjects eligible for inclusion in the Core Phase of the study fulfilled the following key inclusion criteria:

* Subject was an adult male or female ≥ 18 years of age.
* Subjects with histologically and/or cytologically confirmed diagnosis of estrogen receptor (ER)-positive and/or progesterone receptor (PgR)-positive breast cancer by local laboratory.
* Subjects with a confirmed human epidermal growth factor receptor-2 (HER2)-negative aBC.
* Subjects with gene encoding the p110alpha catalytic subunit of PI3K (phosphatidylinositol-3-kinase) (PIK3CA) mutation.
* In case of women, both premenopausal and postmenopausal subjects were allowed to be included in this study.
* Subjects with documented evidence of tumor progression on or after:

  i. Cyclin-Dependent Kinase 4 and 6 inhibitor (CDK4/6i) treatment as last treatment regimen in Cohorts A and B.

ii. aromatase inhibitor (AI) treatment (either in adjuvant or metastatic setting) and received systemic chemotherapy or ET (monotherapy or combination except CDK4/6i + AI) as last treatment regimen in Cohort C. Upon completion of enrollment of Cohort B, subjects who received CDK4/6i + fulvestrant as immediate prior therapy were eligible for Cohort C.

iii. No more than 2 prior anticancer therapies for aBC. iv. Received no more than 1 prior regimen of chemotherapy for the treatment of advanced/metastatic disease was permitted.

v. Recovered to grade 1 or better from any adverse events (AEs) related to previous anticancer therapy prior to study entry (except alopecia or other toxicities not considered a safety risk for the subject at the investigator's discretion).

* Subjects with:

  i. Measurable disease, i.e., at least 1 measurable lesion as per RECIST v1.1 criteria; or ii. If no measurable disease was present, at least 1 predominantly lytic bone lesion had to be present.
* Subjects with adequate bone marrow and coagulation function, liver function and renal function as shown by laboratory values.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.

Key exclusion criteria were:

* Subjects with a known hypersensitivity to alpelisib, fulvestrant, letrozole, goserelin, or leuprolide or to any of their excipients.
* Subjects with prior treatment with any PI3K inhibitor (PI3Ki).
* Subjects with central nervous system (CNS) involvement unless they met all of the following criteria:

  i. At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment, ii. Clinically stable CNS tumor at the time of screening untreated or without evidence of progressions for at least 4 weeks after treatment as determined by clinical examination and brain imaging (magnetic resonance imaging (MRI) or computed tomography (CT) during screening period and stable low dose of steroids for 2 weeks prior to initiating study treatment.
* Subjects with an established diagnosis of diabetes mellitus type I or uncontrolled type II.
* Any concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate subject participation in the study (e.g., chronic active hepatitis, severe hepatic impairment, etc.).
* Subjects with a history of noncompliance to medical regimens.
* Subjects with impairment of gastrointestinal (GI) function or GI disease that could significantly alter the absorption of the study drugs based on investigator discretion.
* Subjects with documented pneumonitis/interstitial lung disease which was active and requiring treatment.
* Subjects concurrently using other anticancer therapy. All anticancer therapy had to be discontinued prior to Day 1 of study treatment.
* Subjects who had major surgery within 14 days prior to starting treatment with alpelisib, or did not recover from major side effects.
* Subjects with significant cardiac abnormalities.
* History of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis.
* Subjects who did not use highly effective contraception while on alpelisib and through the duration after the final dose of alpelisib (not applicable to postmenopausal women).
* Subjects with unresolved osteonecrosis of the jaw.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (88):
- United States (25):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Kaiser Permanente Medical Group, Anaheim, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of Calif Irvine Med Cntr, Irvine, California
  - Kaiser Permanent Southern Californi, San Diego, California
  - UCSF, San Francisco, California
  - Yale University Yale Cancer Center, New Haven, Connecticut
  - Advent Health Cancer Institute, Orlando, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Med Center Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Josephine Ford Cancer Center, Detroit, Michigan
  - St Vincent Frontier Cancer Center, Billings, Montana
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Memorial Sloane Ketterin Cancer Ctr, New York, New York
  - Uni Hosp of Cleveland Cancer Center, Cleveland, Ohio
  - Texas Oncology, Dallas, Texas
  - Cancer Care Centers of South Texas HOAST, San Antonio, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Medical Specialists, Tacoma, Washington
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, La Rioja
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Chile (2):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Santiago
- Denmark (2):
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Vejle
- France (10):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Delhi, India
- Israel (4):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Osaka, Osaka, Japan
- Novartis Investigative Site, Jalisco, Mexico
- Novartis Investigative Site, Maastricht, Limburg, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Castellon
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- United Kingdom (5):
  - Novartis Investigative Site, Edinburgh, Scotland
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rugo HS, Lerebours F, Ciruelos E, Drullinsky P, Ruiz-Borrego M, Neven P, Park YH, Prat A, Bachelot T, Juric D, Turner N, Sophos N, Zarate JP, Arce C, Shen YM, Turner S, Kanakamedala H, Hsu WC, Chia S. Alpelisib plus fulvestrant in PIK3CA-mutated, hormone receptor-positive advanced breast cancer after a CDK4/6 inhibitor (BYLieve): one cohort of a phase 2, multicentre, open-label, non-comparative study. Lancet Oncol. 2024 Dec;25(12):e629-e638. doi: 10.1016/S1470-2045(24)00673-9. PMID 39637900
- [Derived] Borrego MR, Lu YS, Reyes-Cosmelli F, Park YH, Yamashita T, Chiu J, Airoldi M, Turner N, Fein L, Ghaznawi F, Singh J, Pantoja K, Schnell C, Akdere M, Chia S. SGLT2 inhibition improves PI3Kalpha inhibitor-induced hyperglycemia: findings from preclinical animal models and from patients in the BYLieve and SOLAR-1 trials. Breast Cancer Res Treat. 2024 Nov;208(1):111-121. doi: 10.1007/s10549-024-07405-8. Epub 2024 Aug 23. PMID 39177931
- [Derived] Rodon J, Demanse D, Rugo HS, Burris HA, Simo R, Farooki A, Wellons MF, Andre F, Hu H, Vuina D, Quadt C, Juric D. A risk analysis of alpelisib-induced hyperglycemia in patients with advanced solid tumors and breast cancer. Breast Cancer Res. 2024 Mar 4;26(1):36. doi: 10.1186/s13058-024-01773-1. PMID 38439079
- [Derived] Rugo HS, Lerebours F, Ciruelos E, Drullinsky P, Ruiz-Borrego M, Neven P, Park YH, Prat A, Bachelot T, Juric D, Turner N, Sophos N, Zarate JP, Arce C, Shen YM, Turner S, Kanakamedala H, Hsu WC, Chia S. Alpelisib plus fulvestrant in PIK3CA-mutated, hormone receptor-positive advanced breast cancer after a CDK4/6 inhibitor (BYLieve): one cohort of a phase 2, multicentre, open-label, non-comparative study. Lancet Oncol. 2021 Apr;22(4):489-498. doi: 10.1016/S1470-2045(21)00034-6. PMID 33794206
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 92 centers across 19 countries
Pre-assignment Details: Screening assessments occurred before 21 days of the start of treatment.
Groups:
- Cohort A: Pre-treated With CDK 4/6i + AI: Participants who received any CDK 4/6i plus AI as immediate prior treatment will receive alpelisib + fulvestrant
Period: Core Phase
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Started | 127 | 126 | 126
Completed | 1 | 0 | 10
Not Completed | 126 | 126 | 116
Not completed — Progressive disease | 89 | 88 | 90
Not completed — Adverse Event | 20 | 14 | 13
Not completed — Physician Decision | 7 | 13 | 5
Not completed — Subject/guardian decision | 5 | 8 | 4
Not completed — Death | 3 | 2 | 4
Not completed — Protocol deviation | 1 | 1 | 0
Not completed — Technical problems | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Started | 1 | 0 | 10
Completed | 0 | 0 | 5
Not Completed | 1 | 0 | 5
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Subject/guardian decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort C: Pre-treated With Systemic Chemotherapy or ET: Participants who received systemic chemotherapy or ET (as monotherapy or in combination with targeted treatment except CDK 4/6i + AI) as immediate prior treatment will receive alpelisib + fulvestrant.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET | Total
Number analyzed (Participants) | 127 | 126 | 126 | 379
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 80 | 83 | 258
  >=65 years | 32 | 46 | 43 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 126 | 125 | 378
  Male | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 81 | 85 | 83 | 249
  Unknown | 23 | 24 | 11 | 58
  Asian | 12 | 8 | 28 | 48
  Black | 6 | 1 | 1 | 8
  Other | 3 | 7 | 3 | 13
  Pacific islander | 1 | 0 | 0 | 1
  Missing | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Percentage of Participants Who Were Alive Without Disease Progression at 6 Months
Description: Percentage of participants who were alive without disease progression at 6-month follow-up based on local investigator assessment per RECIST v1.1 in Cohort A, Cohort B and Cohort C. Participants who progressed, died, or discontinued study before 6 months were counted as a failure.
Time Frame: At 6 months
Population: Subjects who have been assigned and received at least one dose of the study treatment. They must have a confirmed PI3KCA mutation from a Novartis designated laboratory.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Percentage of participants | 53.8 [44.41 to 62.96] | 46.5 [37.10 to 56.07] | 53.0 [43.51 to 62.41]

2. Secondary Outcome: Core Phase: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study medication to the date of the first documented progression or death due to any cause occurring in the study. PFS was assessed based on local investigator's assessment according to RECIST v1.1. PFS was censored if no PFS event was observed before the cut-off date. The censoring date was the date of last adequate tumor assessment before the cut-off date. If a PFS event was observed after two or more missing or non-adequate tumor assessments, then PFS was censored at the last adequate tumor assessment. PFS was estimated using the Kaplan-Meier method.
Time Frame: From date of first dose to date of first documented progression or death, up to 46 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Months | 8.0 [5.6 to 8.6] | 5.6 [3.7 to 7.1] | 5.6 [5.4 to 8.1]

3. Secondary Outcome: Core Phase: Progression Free Survival on Next Line Treatment (PFS2)
Description: PFS2 is defined as time from the date of first dose of study medication to the date of first documented progression on next-line therapy or death from any cause. The first documented progression on next-line treatment is based on investigator assessment of progressive disease. PFS2 was estimated using the Kaplan-Meier method.
Time Frame: From date of first dose to date of first documented progression on next-line therapy or death, up to approximately 55 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Months | 15.2 [11.4 to 21.7] | 13.0 [10.2 to 13.9] | 13.5 [11.5 to 17.3]

4. Secondary Outcome: Core Phase: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST v1.1 in each cohort. CR: Disappearance of all non-nodal target lesions and all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm and all lymph nodes assigned as non-target lesions must be non-pathological in size (<10 mm short axis) PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 46 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Percentage of participants | 19.3 [12.7 to 27.6] | 17.5 [11.1 to 25.8] | 25.2 [17.6 to 34.2]

5. Secondary Outcome: Core Phase: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with a BOR of CR or PR or an overall lesion response of stable disease (SD) or Non-CR/ Non-PD lasting ≥ 24 weeks based on local investigator's assessment according to RECIST v1.1. CR: Disappearance of all non-nodal target lesions and all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm and all lymph nodes assigned as non-target lesions must be non-pathological in size (<10 mm short axis) PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to 46 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Percentage of participants | 46.2 [37.0 to 55.6] | 35.1 [26.4 to 44.6] | 38.3 [29.4 to 47.8]

6. Secondary Outcome: Core Phase: Duration of Response (DOR)
Description: DOR is the time from the date of first documented response (confirmed CR or PR based on local investigator's assessment according to RECIST v1.1) to the date of first documented progression or death due to underlying cancer. Subjects continuing without progression or death due to underlying cancer were censored at the date of their last adequate tumor assessment. DOR was estimated using the Kaplan-Meier method.
Time Frame: From date of first documented response to first documented progression or death, up to 33.3 months
Population: Subjects who have been assigned and received at least one dose of the study treatment. They must have a confirmed PI3KCA mutation from a Novartis designated laboratory. Additionally, subjects must have a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 23 | 20 | 29
Months | 13.8 [5.5 to 19.4] | 6.5 [5.4 to 9.4] | 16.5 [8.3 to 22.2]

7. Secondary Outcome: Core Phase: Overall Survival (OS)
Description: OS is defined as the time of start of treatment to date of death or lost to follow-up. If a subject was not known to have died, then the OS data was censored at the date of the last known alive status for the patient.
Time Frame: From date of first dose and up to approximately 55 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant | Cohort C: Pre-treated With Systemic Chemotherapy or ET
Number analyzed (Participants) | 119 | 114 | 115
Months | 27.3 [21.3 to 32.7] | 29.0 [24.5 to 34.8] | 20.7 [16.9 to 28.1]

8. Secondary Outcome: Extension Phase: Percentage of Participants With Clinical Benefit as Assessed by the Investigator During the Extension Phase
Description: Clinical Benefit Rate, as assessed by the Investigator during the Extension Phase, was defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR), or an overall lesion response of Stable Disease (SD) or non-complete response/non-progressive disease that lasted at least 24 weeks, based on the local investigator's assessment according to Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: Day 1 of each extension cycle up to Cycle 29 (each cycle lasting 28 days); median duration of exposure to study treatment (alpelisib or fulvestrant) = 41 months
Population: All subjects in Extension Phase who received at least 1 dose of study treatment. All patients consisted of 1 patient from Cohort A and 10 patients from Cohort C pulled together.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients in Extension Phase: Patients with clinical benefit in Extension Phase
Arm/Group | All Patients in Extension Phase
Number analyzed (Participants) | 11
Participants
  Extension Cycle 1 Day 1 | 8
  Extension Cycle 2 Day 1 | 7
  Extension Cycle 3 Day 1 | 7
  Extension Cycle 4 Day 1 | 6
  Extension Cycle 5 Day 1 | 8
  Extension Cycle 6 Day 1 | 7
  Extension Cycle 7 Day 1 | 7
  Extension Cycle 8 Day 1 | 6
  Extension Cycle 9 Day 1 | 7
  Extension Cycle 10 Day 1 | 5
  Extension Cycle 11 Day 1 | 4
  Extension Cycle 12 Day 1 | 7
  Extension Cycle 13 Day 1 | 4
  Extension Cycle 14 Day 1 | 5
  Extension Cycle 15 Day 1 | 4
  Extension Cycle 16 Day 1 | 3
  Extension Cycle 17 Day 1 | 3
  Extension Cycle 18 Day 1 | 3
  Extension Cycle 19 Day 1 | 3
  Extension Cycle 20 Day 1 | 3
  Extension Cycle 21 Day 1 | 3
  Extension Cycle 22 Day 1 | 3
  Extension Cycle 23 Day 1 | 3
  Extension Cycle 24 Day 1 | 2
  Extension Cycle 25 Day 1 | 2
  Extension Cycle 26 Day 1 | 2
  Extension Cycle 27 Day 1 | 2
  Extension Cycle 28 Day 1 | 2
  Extension Cycle 29 Day 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the first dose through post-treatment follow-up, for up to 86 months. Deaths were recorded from study start through post-treatment follow-up over the same period. AE data were summarized for core phase patients from start to end of the core phase (up to 58 months) and for extension phase patients from the start of the core phase through the end of the extension phase (up to 86 months).
Description: No patient from Cohort B entered Extension Phase
Groups:
- Cohort A: Pre-treated With CDK 4/6i + AI (Core Phase): Cohort A: Pre-treated with CDK 4/6i + AI (Core Phase) - Events from the start to end of the Core Phase (up to 58 months)
- Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Core Phase): Cohort B: Pre-treated with CDK 4/6i + fulvestrant (Core Phase) - Events from the start to end of the Core Phase (up to 58 months)
- Cohort C: Pre-treated With Systemic Chemotherapy or ET (Core Phase): Cohort C: Pre-treated with systemic chemotherapy or ET (Core Phase) - Events from the start to end of the Core Phase (up to 58 months)
- Cohort A: Pre-treated With CDK 4/6i + AI (Extension Phase): Cohort A: Pre-treated with CDK 4/6i + AI (Extension Phase) - Events from the start of the Core Phase through the end of the Extension Phase (up to 86 months)
- Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Extension Phase): Cohort B: Pre-treated with CDK 4/6i + fulvestrant (Extension Phase) - Events from the start of the Core Phase through the end of the Extension Phase (up to 86 months)
- Cohort C: Pre-treated With Systemic Chemotherapy or ET (Extension Phase): Cohort C: Pre-treated with systemic chemotherapy or ET (Extension Phase) - Events from the start of the Core Phase through the end of the Extension Phase (up to 86 months)
Arm/Group | Cohort A: Pre-treated With CDK 4/6i + AI (Core Phase) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Core Phase) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Core Phase) | Cohort A: Pre-treated With CDK 4/6i + AI (Extension Phase) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Extension Phase) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Extension Phase)
All-Cause Mortality (participants affected / at risk) | 78/127 | 76/126 | 67/126 | 0/1 | 0/0 | 1/10
Serious Adverse Events (participants affected / at risk) | 37/127 | 48/126 | 38/126 | 0/1 | 0/0 | 3/10
Other Adverse Events (participants affected / at risk) | 126/127 | 126/126 | 124/126 | 1/1 | 0/0 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Pre-treated With CDK 4/6i + AI (Core Phase) (N=127) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Core Phase) (N=126) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Core Phase) (N=126) | Cohort A: Pre-treated With CDK 4/6i + AI (Extension Phase) (N=1) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Extension Phase) (N=0) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Extension Phase) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 2 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 3 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Pre-treated With CDK 4/6i + AI (Core Phase) (N=127) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Core Phase) (N=126) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Core Phase) (N=126) | Cohort A: Pre-treated With CDK 4/6i + AI (Extension Phase) (N=1) | Cohort B: Pre-treated With CDK 4/6i + Fulvestrant (Extension Phase) (N=0) | Cohort C: Pre-treated With Systemic Chemotherapy or ET (Extension Phase) (N=10)
Anaemia (Blood and lymphatic system disorders) | 11 | 9 | 9 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 7 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 7 | 6 | 5 | 1 | 0 | 1
Eye oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 3 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 10 | 4 | 6 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 3 | 3 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 17 | 21 | 10 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 16 | 17 | 6 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 12 | 16 | 15 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 82 | 86 | 68 | 1 | 0 | 7
Dry mouth (Gastrointestinal disorders) | 11 | 10 | 11 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 19 | 13 | 13 | 1 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 0 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 59 | 68 | 51 | 1 | 0 | 3
Oral pain (Gastrointestinal disorders) | 2 | 0 | 4 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 34 | 43 | 38 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 31 | 31 | 31 | 0 | 0 | 2
Asthenia (General disorders) | 24 | 27 | 15 | 1 | 0 | 2
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 39 | 38 | 44 | 0 | 0 | 5
Influenza like illness (General disorders) | 5 | 2 | 2 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 5 | 6 | 5 | 0 | 0 | 2
Oedema peripheral (General disorders) | 10 | 12 | 8 | 0 | 0 | 1
Pain (General disorders) | 5 | 3 | 3 | 0 | 0 | 1
Pyrexia (General disorders) | 17 | 19 | 19 | 0 | 0 | 1
Thirst (General disorders) | 2 | 2 | 3 | 0 | 0 | 1
Xerosis (General disorders) | 2 | 2 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 4 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 3 | 1 | 5 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 1 | 2 | 7 | 0 | 0 | 3
Cystitis (Infections and infestations) | 4 | 3 | 4 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 3 | 1 | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 4 | 3 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 3 | 2 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 14 | 11 | 15 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin graft failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 13 | 13 | 18 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 17 | 11 | 15 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 7 | 3 | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 1 | 2 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 3 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 15 | 12 | 8 | 1 | 0 | 2
Blood glucose increased (Investigations) | 2 | 1 | 3 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 2
Eosinophil count increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 7 | 7 | 2 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 3 | 8 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 2 | 4 | 1 | 0 | 0
Weight decreased (Investigations) | 18 | 19 | 23 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 37 | 56 | 42 | 0 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 76 | 81 | 85 | 1 | 0 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 5 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 12 | 8 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 3 | 1 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 4 | 3 | 5 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21 | 14 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 14 | 12 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 8 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 15 | 14 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 6 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 5 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7 | 7 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 8 | 9 | 7 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 18 | 21 | 8 | 1 | 0 | 1
Headache (Nervous system disorders) | 28 | 25 | 21 | 0 | 0 | 4
Lethargy (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 3 | 0 | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 6 | 3 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 3 | 9 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 4 | 2 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 2 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 1 | 2 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 13 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 14 | 7 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 7 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 20 | 19 | 0 | 0 | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 24 | 16 | 1 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 9 | 7 | 1 | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 0 | 0 | 2
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 1 | 3 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 13 | 29 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 39 | 39 | 51 | 1 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 20 | 9 | 1 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1 | 5 | 0 | 0 | 2
Capillary fragility (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 9 | 11 | 8 | 1 | 0 | 2
Lymphoedema (Vascular disorders) | 2 | 2 | 3 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03056755/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03056755/SAP_002.pdf